CLINICAL TRIAL: NCT05575882
Title: Anti-relapse Efficacy and Tolerance Assessment of a Cosmetic Cream Intended for Very Dry, Irritated to Atopic Sensitive Skin
Brief Title: Anti-relapse Efficacy and Tolerance Assessment of a Cosmetic Cream for Very Dry, Irritated to Atopic Sensitive Skin.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NAOS Argentina S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC2022/PSagc/SG-AR
Record Dates: First submitted 2022-09-27; First posted 2022-10-12 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis; Eczema, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Multicentric, double blind, randomized, comparative study with two parallel group: study group vs placebo group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: white plastic bottles and automatized randomization in eCRF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational product (BI 479 V1) (Active Comparator): The study product or placebo will be applied twice daily on a clean and dry skin for 120 days. Follow "3-6-9 method" as follows: for babies (6 months to 24 months) use 3 pumps for the whole body (1 pump for face, 1 pump for trunk and arms and 1 pump for lower limbs), for children from 25 months: use 6 pumps for the whole body (1 pump for face, 3 pumps for trunk and arms and 2 pumps for lower limbs) and for children with height greater than 1.5 meters: use 9 pumps for the whole body (1 pump for face, 1 pump for chest, 1 pump for back, 1 pump per arm (x2) and 2 pumps per leg (x2). It will be applied from inclusion visit simultaneously with topical treatment in the following order: first the study product or placebo on the whole body followed by the topical treatment on the flare-up areas.
  Interventions: Other: Skin hydration; Other: Barrier function measurement; Other: Potential of hydrogen measurement (pH); Other: Clinical evaluation of atopic dermatitis; Other: Quality of life assessment; Other: Assessment of the effect on itching and sleep disturbances; Other: Assessment of the tolerance of the study product or placebo
- Placebo (BI 006) (Placebo Comparator): Same instructions of use as active comparator.
  Interventions: Other: Skin hydration; Other: Barrier function measurement; Other: Potential of hydrogen measurement (pH); Other: Clinical evaluation of atopic dermatitis; Other: Quality of life assessment; Other: Assessment of the effect on itching and sleep disturbances; Other: Assessment of the tolerance of the study product or placebo

INTERVENTIONS:
Other: Skin hydration — Skin hydration outside flare-up areas on an initial dry skin (the same in each visit). Non invasive technique.
  Other Names: Corneometer
Other: Barrier function measurement — TEWL measurement outside flare-up areas on an initial dry skin (the same in each visit). Non invasive technique.
  Other Names: Transepidermal Water Loss (TEWL)
Other: Potential of hydrogen measurement (pH) — pH measurement outside flare-up areas on an initial dry skin (the same in each visit). Non invasive technique.
Other: Clinical evaluation of atopic dermatitis — EASI score on each visit. Non invasive technique.
  Other Names: Eczema Area and Severity Index (EASI)
Other: Quality of life assessment — Cardiff questionnaires to assess quality of life of subjects and their family members.
Other: Assessment of the effect on itching and sleep disturbances — Visual analogue scale from 0 to 10
Other: Assessment of the tolerance of the study product or placebo — By collection of Adverse Events (AEs) on daily log and electronic Case Report Form (eCRF).

SUMMARY:
Multicentric, double blind, randomized, comparative study with two parallel group: study group vs placebo group. 5 visits: inclusion visit [day (D) 0] and 4 follow-up visits (D30, D60, D90, and D120).

DETAILED DESCRIPTION:
This is a prospective, double blind, multicentric and comparative study including 5 visits (on D0 which corresponds to inclusion visit, D30, D60, D90, and D120). It will take place from June 2024 to June 2025 in Argentina (CIREC LATAM, Buenos Aires) and India (CIDP, New Dheli). This study will include 100 patients (50 in India and 50 in Argentina) who will be followed up for 120 days (± 3 days).

ELIGIBILITY:
Inclusion Criteria:

* General criteria:

Healthy subject (except AD and other atopic diseases - allergic rhinitis, conjunctivitis, and asthma). The subject can keep its usual treatment (antihistamines, inhaled corticosteroids, and antileukotriene treatment) during the study if applicable. Written informed consent from the subject's parent(s)/legal representative(s) and children over 8 years old (specific Argentina) and over 12 years old (specific Singapore). Subject accepting to continue the normal conditions of hygiene and sunscreen (if applicable). Subject, parents/legal representative(s) willing to adhere to the study protocol and procedures.

Specific criteria:

Sex: male or female. Age: from 6 months to 15 years. Subject having on average one flare-up per month during the four months preceding the study, including the one observed on the inclusion visit D0. Subject having EASI value from 7.1 - 21 on D0 (moderate AD). Subject having one atopic eruption on the inclusion visit which the dermatologist will prescribe topical corticosteroids or calcineurin's inhibitors (pimecrolimus and/or tacrolimus).

Exclusion Criteria:

* Subject presenting cutaneous pathology in the studied zone other than AD (according to the investigator's appreciation, i.e., acne, psoriasis). Subject using systemic treatment, including oral steroids and oral immunosuppressants e.g., ciclosporin during the previous weeks liable to interfere with the assessment of the cutaneous tolerance of the study product or placebo (according to the investigator's appreciation). Subject using skin-moisturizing products from inclusion (D0) other than the study product or placebo. Subject who had systemic therapy with immune-suppressive drugs and antibiotics within the last 14 days before the beginning of the study Subject having serious illness that might require regular systemic medication (e.g., insulin-dependent diabetes, cancer) or conditions that exclude a participation or might influence the study evaluation. Subject with documented allergies to the study product or placebo ingredients. Subject enrolled in another clinical study during the study period. Parent(s)/legal representative(s) considered by the investigator to be likely not compliant to the protocol.

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change of acute flares of eczema in patients with chronic atopic dermatitis (AD) | 4 months
  Clinical evaluation by dermatologist on each visit and daily log statements by the parents.

SECONDARY OUTCOMES:
Change of Atopic Dermatitis using the Eczema Area and Severity Index (EASI) | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Clinical evaluation by dermatologist on each visit. Minimum value: 0; maximum value:72. Higher scores mean worse outcome.
Change of Atopic Dermatitis using the Investigator's Global Assessment (IGA) | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Clinical evaluation by dermatologist on each visit. Minimum value: 0; maximum value:4. Higher scores mean worse outcome.
Tolerance of the study product or placebo | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Collection of treatment-related adverse events during the study
Change of stratum corneum (SC) hydration. | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Measurement performed with -Corneometer® CM825 (Courage + Khazaka) and MPACT + software (Monaderm). Subjects must not have applied anything to the forearms on the morning of the measurements. Subject acclimatize for at least 15 minutes in the lab under standardised conditions, with bare test area: - room temperature: 20-22°C;
  - relative humidity: 40-60%. Dry skin area (the same in all visits): the most recommended area are the forearms (avoid flare-up areas). Minimum value: 0; maximum value:60. Higher scores mean better outcome.
Change on the trans-epidermal water loss (TEWL). | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Measurement performs with - Tewameter® TM Hex (Courage & Khazaka) and MPACT + software (Monaderm). Subjects must not have applied anything to the forearms on the morning of the measurements. Subject acclimatize for at least 15 minutes in the lab under standardised conditions, with bare test area: - room temperature: 20-22°C;
  - relative humidity: 40-60%. Dry skin area (the same in all visits): the most recommended area are the forearms (avoid flare-up areas). Minimum value: 0; maximum value:20. Higher scores mean worse outcome.
Change on the pH. | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Measurement perform with LAQUA pHmeter PHD72G. Subject must not have applied anything to the forearms on the morning of the measurements. Subject acclimatize for at least 15 minutes in the lab under standardised conditions, with bare test area: - room temperature: 20-22°C;
  - relative humidity: 40-60%. Dry skin area (the same in all visits): the most recommended area are the forearms (avoid flare-up areas). Minimum value: 0; maximum value:14. pH higher than 5,9 or lower than 4,5 scores mean worse outcome.
Change on itching | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Interview by dermatologist on each visit. Minimum value: 0; maximum value:10. Higher scores mean worse outcome.
Change on sleep disturbances. | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Interview by dermatologist on each visit. Minimum value: 0; maximum value:10. Higher scores mean worse outcome.
Change on quality of life. | 0-30, 31-60, 61-90 and 91-120 days of treatment
  Cardiff quality of life questionnaires fill in by subjects or parents according to age range. The total score is calculated by summing the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The questionnaires can also be expressed as a percentage of the maximum possible score of 30.
Subjective appreciation of efficacy and acceptability by the parent(s)/legal representative(s) and/or their child. | 120 days
  Questionnaire fill in by representative(s) and/or their child. Score from "totally agree" to "totally disagree". "Totally agree" and "agree" are considered positive answers (in percentage). Somewhat agree and and totally disagree are considered negative answers (in percentage). The questionnaires are expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (3):
- Cirec Latam, Ciudad Autónoma de Buenos Aire, Ciudad Autónoma de Buenos Aire, Argentina
- CIDP, New Delhi, India
- KK Women's & Children's Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gayraud F, Sayag M, Jourdan E. Efficacy and tolerance assessment of a new type of dermocosmetic in infants and children with moderate atopic dermatitis. J Cosmet Dermatol. 2015 Jun;14(2):107-12. doi: 10.1111/jocd.12145. Epub 2015 Mar 23. PMID 25807867